CLINICAL TRIAL: NCT03413293
Title: Nosocomial Bacterial and Fungal Chest Infections in Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, NZBakhiet, resident doctor, Assiut University
Other Study IDs: NBFCIIHCP
Record Dates: First submitted 2018-01-08; First posted 2018-01-29 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-02

CONDITIONS: Nosocomial Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nosocomial infected cirrhotic patients
  Interventions: Diagnostic Test: Diagnosis of bacterial infections

INTERVENTIONS:
Diagnostic Test: Diagnosis of bacterial infections — Cultures

SUMMARY:
Hospital acquired chest Infections are common complications in hospitalized cirrhotic patients. Infectious complications are the most common cause of mortality in cirrhotic patients with bronchopneumonia early antibiotic treatment at the base of culture and sensitivity is an optimal therapeutic approach in cirrhotics with nosocomial pneumonia Intensive care unit acquired pneumonia is the leading infection in critically ill patients and a major cause of morbidity and mortality despite recent major advances in antimicrobial therapy, supportive care, and the use of a broad range of preventive measures

DETAILED DESCRIPTION:
Aim of the work

1. To estimate the frequency and risk factors of nosocomial chest infections in cirrhotic patients .
2. To determine the causative pathogens of nosocomial chest infections in patients with cirrhosis including fungal infections in order to establish our local empirical antimicrobial protocol.
3. To define the impact of nosocomial chest infections on survival of our patients.
4. To develop an effective and continuous surveillance program and infection control measures to reduce the burden of these infections as well as morbidity , mortality , hospital stay ,hospital cost and to achieve quality of care .
5. To motivate pharmaceutical companies to create a new umbrella coverage of antimicrobials through the ongoing knowledge of the changes in microbial resistance pattern inside hospitals

ELIGIBILITY:
Inclusion Criteria:

* All cirrhotic patients , decompensated , child pug score B or C ,may have Hepatocellular carcinoma , other comorbidities may present as (Diabetius mellitus , Hypertension , Heart disease and renal impairment ) , both sex and with clinical suspicion of chest infections acquired after 48 hours of admission

Exclusion Criteria:

* Patients have any chronic chest disease
* Patients have severe immunosuppression (neutropenia after chemotherapy or hematopoietic transplant, drug-induced immunosuppression in solid-organ transplant or cytotoxic therapy, and HIV-related disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient were known to have liver cirrhois and admitted at hospital secondary to any cause
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of nosocomial infection in patients with liver cirrhosis | baseline
  nosocomial infection is one of predictors of bad outcome in liver cirrhosis

REFERENCES:
- [Background] Di Pasquale M, Esperatti M, Crisafulli E, Ferrer M, Bassi GL, Rinaudo M, Escorsell A, Fernandez J, Mas A, Blasi F, Torres A. Impact of chronic liver disease in intensive care unit acquired pneumonia: a prospective study. Intensive Care Med. 2013 Oct;39(10):1776-84. doi: 10.1007/s00134-013-3025-6. Epub 2013 Aug 2. PMID 23907496